CLINICAL TRIAL: NCT00309296
Title: Longitudinal Care: Smoking Reduction to Aid Cessation; Part of Hatsukami's Tobacco Exposure Reduction
Brief Title: Longitudinal Care: Smoking Reduction to Aid Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health (NIH) (NIH)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Anne Joseph, MD, MPH, University of Minnesota
Organization: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TLC; P50DA013333-07 (NIH)
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Diseases
Keywords: smoking cessation; smoking reduction; nicotine replacement therapy
MeSH Terms: conditions — Chronic Disease; Smoking Cessation; Smoking Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Longitudinal Care (Experimental): One year of combined behavioral and pharamcological tobacco dependence treatment, with interim smoking reduciton for smokers who fail initial quit attempt.
  Interventions: Behavioral: smoking cessation
- Usual Care (Active Comparator): Evidence based, state-of-the-science tobacco treatment; combined behavioral and pharmacological treatment for 8 weeks
  Interventions: Behavioral: smoking cessation

INTERVENTIONS:
Behavioral: smoking cessation — This was a randomized controlled trial to compare long-term smoking cessation outcomes between Longitudinal Care (LC) and Usual Care (UC) treatment groups. The LC group received smoking cessation treatment (combined behavioral and pharmacological therapies) for one-year period. This treatment recommended repeat quit attempts or smoking reduction for those who failed to quit after the initial attempt. The UC group received evidence-based treatment that lasted 8 weeks.

SUMMARY:
The purpose of this study is to determine whether an extended care treatment model lasting over a year will increase long-term smoking cessation rates compared to the standard 8 week treatment of care.

DETAILED DESCRIPTION:
Objective The objective of this project is to conduct a randomized controlled trial to compare 1) an extended quality care smoking cessation treatment delivered over a one-year period (EQC) to 2) quality care smoking cessation treatment delivered over an 8 week period (QC) to determine if EQC improves prolonged smoking abstinence.

Research Design/Methodology 500 smokers who are interested in quitting will be enrolled and randomly assigned to the EQC or QC groups. Both groups will initially receive a state-of-the-science smoking cessation intervention including behavioral and pharmacological components, delivered by a combination of in-person and telephone care. EQC participants who fail to quit, reduce but do not quit, or relapse will receive intensive treatment over the ensuing 12 months that encourages repeat quit attempts and smoking reduction if they are not to quit. We propose reduction as an intermediate goal in LC because this may increase the likelihood of cessation, increase self-efficacy and keep smokers and clinicians engaged. Reduction treatment will include behavioral treatment and nicotine replacement. QC participants will only receive occasional prompts to quit. The primary endpoint will be 6M of abstinence measured 18M after enrollment. Secondary endpoints will include point prevalent abstinence, smoking reduction, self-efficacy and satisfaction. We will also collect qualitative data from successful abstainers and reducers about decision making processes and intervention experiences.

Clinical Significance This project will address the potential role of smoking reduction in the treatment menu for smokers interested in quitting. This project examines mechanisms, methods and a "real world" application for reducing toxin exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Current and regular smoker 5 or more cigarettes per day
* Interested in making a quit attempt in the next 14 days
* Personal phone available

Exclusion Criteria:

* Pregnancy or plans to become pregnant in the next year
* Cannot speak English
* Not a union member or employee of specified worksite or immediate family member
* Member of household is currently enrolled in the study
* Not willing to comply with study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be 6M of abstinence measured 18M after enrollment. | 18M
  6M prolonged abstinence

SECONDARY OUTCOMES:
7d point prevalent abstinence | 18M
  Data collected at 21d, 3, 6, 12, 18M
30d point prevalent abstinence | 18M
  Data collected at 3, 6, 12, 18M
Smoking reduction | 18M
  Data collected at 3, 6, 12, 18M
Total duration of abstinence | 18M
  Time Line Follow Back

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Joseph, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- Minneapolis VAMC, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Joseph AM, Fu SS, Lindgren B, Rothman AJ, Kodl M, Lando H, Doyle B, Hatsukami D. Chronic disease management for tobacco dependence: a randomized, controlled trial. Arch Intern Med. 2011 Nov 28;171(21):1894-900. doi: 10.1001/archinternmed.2011.500. PMID 22123795